CLINICAL TRIAL: NCT04962464
Title: The Impact of Fasting Mimicking Diet Program and Calorie Mimetic Supplements on Epigenetic Aging
Brief Title: The Impact of a Fast Diet and Calorie Mimetic Supplements on Epigenetic Aging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: L-Nutra Inc (Industry); Peak Human Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TD-EA-001
Record Dates: First submitted 2021-06-16; First posted 2021-07-15 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: prospective, randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fasting Mimicking Diet + Supplement / Usual Routine (Experimental): Participants in will be asked to begin the Peak Human Labs calorie mimetic supplement. They will also begin on day 1 the 5 day Fasting Mimicking Diet Program. Participants will continue the supplementation for the 90 days and repeat the 5 day Fasting Mimicking Diet Program on days 1, 29 and 57. Starting at day 91, they will return to their usual daily routine.
  Interventions: Dietary Supplement: Peak Human Labs calorie mimetic supplement; Behavioral: Fasting Mimicking Diet
- Supplement / Usual Routine (Experimental): Participants will be asked to begin the Peak Human Labs calorie mimetic supplement. Participants will continue the supplementation for 90 days. Starting at day 91, they will return to their usual daily routine.
  Interventions: Dietary Supplement: Peak Human Labs calorie mimetic supplement
- Usual Routine / Fasting Mimicking Diet + Supplement (Experimental): Participants will have no intervention for the first 90 days, during which they will be asked not to start a new fasting program supplement. At day 91, they will begin the 5-day Fasting Mimicking Diet Program and start the Peak Human Labs calorie mimetic supplement. Participants will continue the supplementation for 90 days and repeat the 5-day Fasting Mimicking Diet Program on days 91, 120, and 148.
  Interventions: Dietary Supplement: Peak Human Labs calorie mimetic supplement; Behavioral: Fasting Mimicking Diet
- Usual Routine / Supplement (Experimental): Participants will have no intervention for the first 90 days, during which they will be asked not to start a new fasting program supplement. At day 91,start the Peak Human Labs calorie mimetic supplement. Participants will continue the supplementation for 90 days.
  Interventions: Dietary Supplement: Peak Human Labs calorie mimetic supplement

INTERVENTIONS:
Dietary Supplement: Peak Human Labs calorie mimetic supplement — Supplement
Behavioral: Fasting Mimicking Diet — Diet
  Arms: Fasting Mimicking Diet + Supplement / Usual Routine; Usual Routine / Fasting Mimicking Diet + Supplement

SUMMARY:
This is a prospective randomized clinical study of 50 patients to evaluate the fasting mimicking diet program by Prolon with a calorie mimetic supplement from Peak Human Labs. This study will be evaluating the effectiveness of the combined intervention over a three month program.

The study will assess the effects that the program has on the participants' biological aging.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age > 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Epigenetic Age Biomarkers | Change from baseline to 3 months
  Outcome epigenetic age testing will test methylation at 850,000 spots on the DNA/
Epigenetic Age Biomarkers | Change from baseline to 6 months
  Outcome epigenetic age testing will test methylation at 850,000 spots on the DNA/

SECONDARY OUTCOMES:
Body Mass Index | Change from baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peak Human Labs, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amano H, Chaudhury A, Rodriguez-Aguayo C, Lu L, Akhanov V, Catic A, Popov YV, Verdin E, Johnson H, Stossi F, Sinclair DA, Nakamaru-Ogiso E, Lopez-Berestein G, Chang JT, Neilson JR, Meeker A, Finegold M, Baur JA, Sahin E. Telomere Dysfunction Induces Sirtuin Repression that Drives Telomere-Dependent Disease. Cell Metab. 2019 Jun 4;29(6):1274-1290.e9. doi: 10.1016/j.cmet.2019.03.001. Epub 2019 Mar 28. PMID 30930169
- [Background] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Background] Chen J, Li Y, Zhu Q, Li T, Lu H, Wei N, Huang Y, Shi R, Ma X, Wang X, Sheng J. Anti-skin-aging effect of epigallocatechin gallate by regulating epidermal growth factor receptor pathway on aging mouse model induced by d-Galactose. Mech Ageing Dev. 2017 Jun;164:1-7. doi: 10.1016/j.mad.2017.03.007. Epub 2017 Mar 24. PMID 28343910